CLINICAL TRIAL: NCT07049822
Title: OPTIMA: Optimising Mammography Assesment Via Blood-based Biomarkers
Brief Title: Optimising Mammography Screening Accuracy With Blood-based Biomarkers
Acronym: OPTIMA
Status: Not yet recruiting | Type: Observational
Sponsor: Vejle Hospital (Other)
Collaborators: Sygehus Lillebaelt (Other)
Responsible Party: Sponsor
Other Study IDs: 24/54432 - OPTIMA
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer screening; blood-based biomarkers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mammography screening positive women: All citizens referred to a clinical mammography at Vejle Hospital or Odense University Hospital in the breast cancer screening program are offered to participate in the study. If the participant agrees, they will have blood drawn and sign a declaration of consent.
  Statistically, approximately 25 % will be diagnosed with breastcancer

SUMMARY:
The project aims to investigate whether breast cancer screening can be improved using blood tests, thereby reducing the number of unnecessary clinical mammographies. The Danish breast cancer screening program was implemented in 2007, and currently, all women aged 50-69 are invited every two years to participate. Those who have a suspecious screening mammography are referred to a clinical mammography where further assesment with more mammographies, ultra-sound and possibly biopsies are conducted. Around 75% of the women that are referred to further assesment can be classified as unnecessary, as no breastcancer is found. This results in avoidable and unpleasant procedures for individuals and strains healthcare resources.

The project seeks to reduce the number of these unnecessary clinical mammographies by investigating whether blood biomarkers can identify women at very low risk of breast cancer after a positive mammography screening. By utilizing blood tests, screening could become more personalized, precise, and resource-efficient for the healthcare system.

DETAILED DESCRIPTION:
The study aims to determine if minor irregularities in blood-based biomarkers can identify women with a very low breast cancer risk. Blood samples will be collected from 1200 women attending clinical mammography/recall after a positive mammography screening. Routine blood analyses will be conducted immediately, while blood for special analyses will be stored at -80 °C until analysis.

The study can be divided into sub-studies:

One that will solely focus on the routine blood analyses and evaluate their potential.

And one that will include the analysis of biomarkers that is not yet incorporated into the routine sample track at Vejle or Odense Hospital to see if the inclusion of special biomarkers can improve the breast cancer risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Danish breast cancer screening program

Exclusion Criteria:

* No clinical mammography conducted

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women referred to a clinical mammography at Vejle Hospital or Odense University Hospital in the breast cancer screening program.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-11-20 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between blood samples and clinical mammography result | 6 weeks from clinical mammography date
  The aim is to investigate the womens chance of being healthy despite a positive tmammography screening. The chance of being healthy is estimated from the combined blood sample results and will be compared to the results of the clinical mammography.

SECONDARY OUTCOMES:
Correlation between blood samples and interval breast cancer | From 6 weeks after the clinical mammography to next mammographyscreening, up to 3 years
  The chance of being healthy is estimated from the combined blood sample results and will be compared to the interval cancers diagnosed in the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jonna S Madsen, Prof., MD, Study Chair — Sygehus Lillebaelt; Sisse H Njor, Professor, Study Chair — Sygehus Lillebaelt
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No
Due to Danish regulations IPD is not allowed to be shared without direct approval from the individual. The outcomes of this study can be explored and presented without requiring IPD .